CLINICAL TRIAL: NCT05949801
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase III Clinical Trial Based on Standard Treatment to Evaluate the Effect of Injectable Neucardin on Cardiac Function and Reverse Ventricular Remodeling in Patients With Chronic Systolic Heart Failure
Brief Title: Evaluation of the Effect of Injectable Neucardin on Cardiac Function and Reversal Ventricular Remodeling in Patients With Chronic Systolic Heart Failure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zensun Sci. & Tech. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZS-01-308B
Record Dates: First submitted 2023-06-02; First posted 2023-07-18 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Chronic Systolic Heart Failure
Keywords: CHF Neucardin
MeSH Terms: interventions — Injections

STUDY DESIGN:
Intervention Model Description: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase III Clinical Trial
Who Masked: Participant, Investigator
Masking Description: This trial is planned to be conducted simultaneously in multiple clinical study sites nationwide, including 198 subjects, 99 subjects in the treatment group and 99 subjects in the placebo group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational drug group (Experimental): Neucardin+standard basic therapeutic medication
  Interventions: Drug: Neucardin
- placebo group (Placebo Comparator): Placebo + standard basic therapeutic medication
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Neucardin — 10 days IV infusion of 0.6 ug/kg/day
  Other Names: Recombinant human Neuregulin-1 for Injection
  Arms: Investigational drug group
Drug: Placebo — 10 days IV infusion of 0 ug/kg/day
  Other Names: Excipients of recombinant human neuregulin-1 freeze dried for injection
  Arms: placebo group

SUMMARY:
A multicenter, randomized, double-blind, placebo-controlled phase III clinical trial to evaluate the effect of recombinant human Neuregulin-1 for injection on cardiac function and reverse ventricular remodeling in male patients with NT-proBNP ≤ 1700 pg/ml and female patients with NT-proBNP ≤ 4000 pg/ml and New York Heart Association class II-III chronic systolic heart failure, and to confirm its efficacy and safety.

DETAILED DESCRIPTION:
This trial is planned to be conducted simultaneously in multiple clinical study sites nationwide, including 198 subjects, 99 subjects in the treatment group and 99 subjects in the placebo group.

Primary endpoint:

1.Response rate at 35 days of simultaneous reduction of LVESVI and LVEDVI by more than or equal to 20 ml/m2 (The proportion of the subjects achieving this criterion in each treatment group.)

Secondary endpoints:

1. Response rate at 35 day of LVESVI improvement greater than or equal to 25 ml/m2 ;
2. Response rate at 35 day of LVEDVI improvement greater than or equal to 25 ml/m2 ;
3. Change from baseline in LVEF, LVESV, LVEDV, LVESVI and LVEDVI at 35 days ;
4. 90-day response rate of LVESVI improved greater than or equal to 25ml/m2,LVEDVI improved greater than or equal to 25 ml/m2, and LVESVI and LVEDVI improved greater than or equal to 20 ml/m2 at the same time ;
5. Change from baseline in LVEF, LVESV, LVEDV, LVESVI and LVEDVI at 90 days ;
6. Change from baseline in NYHA at 35 and 90 days ;
7. Change from baseline in quality of life at 35 and 90 days ;
8. Mortality during the study period.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years, male or female;
2. Definite diagnosis of heart failure for 6 months or more, current stable disease, NYHA class II-III, left ventricular ejection fraction (LVEF) ≤ 40%(echocardiographic modified Simpson's method measurement ≤ 40% at screening, and CMR measurement ≤ 40% at baseline);
3. NT-proBNP ≤1700 pg/ml in males and ≤4000pg/ml in females (detected by Roche kit in central laboratory);
4. Receiving standard basic treatment for heart failure for at least 3 months, and did not change the type and dose of heart failure treatment drugs within 1 month;
5. Understand and sign the informed consent form.

Exclusion Criteria:

1. Unable to receive CMR examination, such as patients with pacemakers, ICDs, CRTs, or other similar devices contraindicated for CMR, claustrophobia, atrial fibrillation during the screening period, or inability to cooperate with air-closed activities required for CMR testing;
2. Hypertrophic cardiomyopathy with left ventricular outflow tract obstruction, constrictive pericarditis, significant and uncorrected valvular heart disease, severe valvular regurgitation or severe stenosis, congenital heart disease requiring surgical treatment but not surgical treatment, primary pulmonary hypertension or secondary severe pulmonary hypertension (≥ 70 mmHg), and right heart failure due to pulmonary disease;
3. Patients suffering from proliferative glands or adenomas with endocrine activity which may affect cardiac function or endocrine function, such as pheochromocytoma, thyromegaly, etc. (patients with euthyroid thyroid nodules do not need to be excluded);
4. LVESVi less than 135 ml/m2 at baseline;
5. Prepare to install pacemaker, ICD, CRT or other similar devices within 6 months;
6. History of heart transplantation, use of ventricular assist devices (VADs) or preparation for heart transplantation, VADs;
7. Diagnosis of peripartum or chemotherapy-induced cardiomyopathy within the past 12 months;
8. Subjects with chronic heart failure with acute hemodynamic disturbance or acute decompensation within the past 1 month (symptoms and signs prove that chronic heart failure is aggravated and intravenous drug therapy is required);
9. Angina pectoris within the past 3 months;
10. Myocardial infarction, cerebrovascular accident, revascularization (PCI or other surgery), cardiac surgery, carotid artery or other large vessel surgery within the past 6 months;
11. Serious ventricular arrhythmias (sustained ventricular tachycardia or other conditions that the investigator considers necessary to exclude);
12. Clinical diagnosis of pericardial effusion, pleural effusion or imaging showed pericardial effusion (greater than 50ml or 3 mm or a small amount or more) or pleural effusion (greater than 200ml or 10 mm);
13. Liver and kidney dysfunction and chronic liver disease may have a potential impact on liver function (such as active chronic hepatitis, etc.), non-heart failure causes of bilirubin or alkaline phosphatase > 2 times the upper limit of normal, aspartate aminotransferase and/or alanine aminotransferase > 3 times the upper limit of normal, eGFR calculated using MDRD method < 30 ml/min/1.73 m2;
14. Systolic blood pressure < 90 mmHg or > 160 mmHg;
15. Serum K + < 3.2 mmol/L or > 5.5 mmol/L;
16. Women of childbearing potential who plan to become pregnant within 2 years (women of childbearing potential are defined as all women with physical ability to become pregnant), pregnant or lactating women;
17. Previous history of cancer or current cancer, or pathological examination confirmed precancerous lesions (Such as ductal carcinoma in situ of the breast, or atypical hyperplasia of the cervix), or through the examination (physical examination, X-ray examination or B ultrasound examination or other means) found in vivo malignant mass subjects;
18. The investigator judges that the survival time is expected to be less than 6 months;
19. Participated in any drug clinical trials within the first 3 months;
20. Severe neurological disease (Alzheimer's disease, progressive parkinsonism);
21. Subjects who are unable to complete this study or fail to comply with the requirements of this study (due to administrative reasons or other reasons), as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2023-04-13 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-10-14 (Actual)

PRIMARY OUTCOMES:
Response rate at 35 days of simultaneous reduction of LVESVI and LVEDVI by more than or equal to 20 ml/m2 (The proportion of the subjects achieving this criterion in each treatment group) | Day 35
  Response rate at 35 days of simultaneous reduction of LVESVI and LVEDVI by more than or equal to 20 ml/m2 (The proportion of the subjects achieving this criterion in each treatment group)

SECONDARY OUTCOMES:
Response rate at 35 day of left ventricular end systolic volume index (LVESVI) improvement greater than or equal to 25 ml/m2; | Day 35
  Response rate at 35 day of LVESVI improvement greater than or equal to 25 ml/m2;
Response rate at 35 day of left ventricular end diastolic volume index (LVEDVI) improvement greater than or equal to 25 ml/m2; | Day 35
  Response rate at 35 day of LVEDVI improvement greater than or equal to 25 ml/m2;
Change from baseline in left ventricular ejection fraction (LVEF) at 35 days; | Day 35
  Change from baseline in LVEF at 35 days;
Change from baseline in left ventricular end systolic volume (LVESV) at 35 days; | Day 35
  Change from baseline in LVESV at 35 days;
Change from baseline in left ventricular end diastolic volume (LVEDV) at 35 days; | Day 35
  Change from baseline in LVEDV at 35 days;
Change from baseline in LVESVI and LVEDVI at 35 days; | Day 35
  Change from baseline in LVESVI and LVEDVI at 35 days;
90-day response rate of LVESVI improved greater than or equal to 25 ml/m2; | Day 90
  90-day response rate of LVESVI improved greater than or equal to 25 ml/m2;
90-day response rate of LVEDVI improved greater than or equal to 25 ml/m2; | Day 90
  90-day response rate of LVEDVI improved greater than or equal to 25 ml/m2;
90-day response rate of LVESVI and LVEDVI improved greater than or equal to 20 ml/m2 at the same time; | Day 90
  90-day response rate of LVESVI and LVEDVI improved greater than or equal to 20 ml/m2 at the same time;
Change from baseline in LVEF at 90 days; | Day 90
  Change from baseline in LVEF at 90 days;
Change from baseline in LVESV at 90 days; | Day 90
  Change from baseline in LVESV at 90 days;
Change from baseline in LVEDV at 90 days; | Day 90
  Change from baseline in LVEDV at 90 days;
Change from baseline in LVESVI and LVEDVI at 90 days; | Day 90
  Change from baseline in LVESVI and LVEDVI at 90 days;
Change from baseline in New York Heart Association (NYHA) at 35 and 90 days; | Day 35 and Day 90
  Change from baseline in NYHA at 35 and 90 days;
Change from baseline in quality of life at 35 and 90 days; | Day 35 and Day 90
  Change from baseline in quality of life at 35 and 90 days;The benefit of patients is reflected by the quality of life score table.
Mortality during the study period; | Through study completion, an estimation of average of 1 year
  Mortality during the study period;

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhang, M.D, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital; Mulei Chen, M.D, Principal Investigator — Beijing Chao Yang Hospital
Locations (103):
- China (103):
  - Beijing Chao-Yang Hospital , Capital Medical University, Beijing, Beijing Municipality
  - Beijing Anzhen Hospital , Capital Medical University, Beijing, Beijing Municipality
  - Beijing Friendship Hospital , Capital Medical University, Beijing, Beijing Municipality
  - Chinese people's liberation army general hospital No.6 medical center, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - The First Medical Center of General Hospital of Chinese People's Liberation Army, Beijing, Beijing Municipality
  - Fuwai Hospital Chinese Academy of Medical Sciences, Beijin, Beijing Municipality
  - Chongqing Emergency Medical Center (Chongqing Fourth People's Hospital), Chongqing, Chongqing Municipality
  - Chongqing University Three Gorges Hospital, Chongqing, Chongqing Municipality
  - Longyan First Hospital, Longyan, Fujian
  - Xiamen Cardiovascular Hospital Xiamen University, Xiamen, Fujian
  - First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Guangdong Jieyang People's Hospital, Jieyang, Guangdong
  - Maoming people's hospital, Maoming, Guangdong
  - Liuzhou worker's hospital, Liuchow, Guangxi
  - People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Haikou People's Hospital, Haikou, Hainan
  - Hainan Provincial People's Hospital, Haikou, Hainan
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Qiqihar first hospital, Qiqihar, Heilongjiang
  - Anyang People's Hospital (Anyang Central Hospital), Anyang, Henan
  - Huaihe Hospital of Henan University, Kaifeng, Henan
  - First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Luoyang Central Hospital, Luoyang, Henan
  - Nanyang Central Hospital, Nanyang, Henan
  - Nanyang First People's Hospital, Nanyang, Henan
  - General Hospital of Puyang Oilfield, Puyang, Henan
  - Sanmenxia Central Hospital, Sanmenxia, Henan
  - First People's Hospital of Shangqiu, Shangqiu, Henan
  - The First Affiliated Hospital of Xinxiang Medical College, Xinxiang, Henan
  - Xinxiang central hospital, Xinxiang, Henan
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The First Affiliated Hospital of Henan University, Zhengzhou, Henan
  - Zhumadian Central Hospital, Zhumadian, Henan
  - Chenzhou First People's Hospital, Chenzhou, Huanan
  - People's Hospital of Wuhan University, Wuhan, Hubei
  - Wuhan Wuchang Hospital, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Xiangyang first people's hospital, Xiangyang, Hubei
  - People's Hospital of Hunan Provincial, Changsha, Hunan
  - South China University Affiliated South China Hospital, Hengyang, Hunan
  - The Second Affiliated Hospital of Nanhua University, Hengyang, Hunan
  - Yueyang Central Hospital, Yueyang, Hunan
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - Changzhou No.2 People's Hospital, Changzhou, Jiansu
  - The First People's Hospital of Changzhou, Changzhou, Jiansu
  - Huai'an First People's Hospital, Huai'an, Jiansu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiansu
  - Zhongda Hospital Southeast University, Nanjing, Jiansu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiansu
  - The Suzhou Municipal Hospital, Suzhou, Jiansu
  - Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiansu
  - Xuzhou Central Hospital, Xuzhou, Jiansu
  - Subei people's hospital, Yangzhou, Jiansu
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - Jilin University Second Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - Ansteel Group Genral Hospital, Anshan, Liaoning
  - Benxi Central Hospital, Benxi, Liaoning
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Zhongshan Hospital Affiliated to Dalian University, Dalian, Liaoning
  - Central Hospital Affiliated to Shenyang Medical College, Shenyang, Liaoning
  - Liaoning Provincial People's Hospital, Shenyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Nanyang Second People's Hospital, Henan, Nanyang
  - Heze Municipal Hospital, Heze, Shandong
  - Jinan Central Hospital, Jinan, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong Province Qianfoshan Hospital, Jinan, Shandong
  - Linyi People's Hospital, Linyi, Shandong
  - Tai'an City Central Hospital, Tai’an, Shandong
  - Zibo Municipal Hospital, Zibo, Shandong
  - Affiliated Hospital of Jining Medical College, Jining, Shangdong
  - Jining first people's hospital, Jining, Shangdong
  - Zaozhuang municipal hospital, Zaozhuang, Shangdong
  - Putuo District Central Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Shanghai Baoshan District Wusong Central Hospital, Shanghai, Shanghai Municipality
  - Shanxi Provincial Cardiovascular Hospital, Taiyuan, Shanxi
  - The First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Affiliated Hospital of Shaanxi University of Traditional Chinese Medicine, Xianyang, Shanxi
  - Xianyang first people's hospital, Xianyang, Shanxi
  - Xianyang Hospital of Yan 'an University, Xianyang, Shanxi
  - The First Affiliated Hospital of Xi 'an Jiaotong University, Xi’an, Shanxi
  - Xi'an Gaoxin Hospital, Xi’an, Shanxi
  - The Fifth People's Hospital of Chengdu, Chengdu, Sichuan
  - Mianyang Central Hospital, Mianyang, Sichuan
  - The First Affiliated Hospital of Dali University, Dali, Yunnan
  - Fuwai Yunnan Cardiovascular Hospital, Kunming, Yunnan
  - The First People's Hospital of Yunnan Province, Kunming, Yunnan
  - The First Affiliated Hospital , Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Affiliated Hospital of Hangzhou Normal University, Hanzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Hanzhou, Zhejiang
  - Jiaxing First Hospital, Jiaxing, Zhejiang
  - Ningbo Huamei Hospital, University of Chinese Academy of Sciences (Ningbo Second Hospital), Ningbo, Zhejiang
  - The First Hospital of Ningbo, Ningbo, Zhejiang
  - First affiliated hospital of Wenzhou medical university, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No
Zensun ensures that the key information about the design of this protocol will be published in a publicly available database such as www.clinicaltrials.gov. After the end of the trial, Zensun will assist the study site to objectively summarize the trial results, use appropriate statistical methods to analyze the trial data, objectively evaluate the safety and efficacy of the drug according to the results, and make a complete written summary report of the clinical trial. Study results will be submitted for publication and/or publication in a publicly available database. If other individuals or institutions related to this study want to publish or publish the study results or related data, they need to obtain the consent of the sponsor in advance. If the sponsor needs to include the name of the investigators in any publication or advertisement, the consent of the investigator should be obtained.